CLINICAL TRIAL: NCT04954989
Title: Phase I Open and Monocentric Clinical Trial With Pharmacokinetic and Pharmacodynamic Determination of Intravenous Recombinant Human Erythropoietin in Male Adults.
Brief Title: Biosimilarity Study of Intravenous Recombinant Human Erythropoietin in Healthy Volunteers
Acronym: RUBI
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Megalabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RUBI
Record Dates: First submitted 2021-06-06; First posted 2021-07-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: reticulocytes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test rHuEpo in a single subcutaneous application. (Experimental): Group T: Test rHuEepo shall be administered subcutaneosly to study participants
  Interventions: Biological: Experimental Erythropoietin subcutaneous injection single dose of 4,000 IU; Biological: Active comparator Erythropoietin subcutaneous injection single dose of 4,000 IU
- Reference rHuEpo in a single subcutaneous application. (Active Comparator): Group T: Reference rHuEepo shall be administered subcutaneosly to study participants
  Interventions: Biological: Experimental Erythropoietin subcutaneous injection single dose of 4,000 IU; Biological: Active comparator Erythropoietin subcutaneous injection single dose of 4,000 IU

INTERVENTIONS:
Biological: Experimental Erythropoietin subcutaneous injection single dose of 4,000 IU — Recombinant Human Erythropoietin: single dose of 4,000 IU (syringe filled with 0.4 mL with 4,000 IU) of the experimental drug should be administered subcutaneously
Biological: Active comparator Erythropoietin subcutaneous injection single dose of 4,000 IU — Recombinant Human Erythropoietin: single dose of 4,000 IU (syringe filled with 0.4 mL with 4,000 IU) should be administered subcutaneously

SUMMARY:
Open label and monocentric Phase I Clinical Trial, to Determine the Pharmacokinetics and Pharmacodynamics of Recombinant Human Erythropoietin for Subcutaneous Use in an Adult Male Population

DETAILED DESCRIPTION:
An open label, balanced, randomized, two treatments, two sequences, two periods, single dose, crossover design will be used to study the pharmacokinetics and pharmacodynamics of two different rHuEpo products when administered subcutaneously in healthy subjects.

PK parameters to evaluate shall be AUCt and AUCt to infinity, and Cmax PD parameter shall be erithrocye and reticulocyte counts and hematocrite. Bioequivalence shall be evaluated according to 80-125 T/R rate for 90 % Cmax and AUC for pk and PD parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy eligible participants able to read, understand and sign the latest version of the Informed Consent Form (FICF) approved by the Research Ethics Committee (CEP);
* Male participants aged between 18 and 55 years;
* Be characterized as a healthy research participant, based on medical history, general physical examination and vital signs, laboratory tests and ECG not indicating any evidence of disease;
* Present BMI ≥ 18 and ≤ 29.9 Kg/m2;
* Have a body weight of 60 - 100 kg;
* Present a negative test for coronavirus.

Exclusion Criteria:

* Present one or more flu-like symptoms such as: fever (body temperature greater than or equal to 37.8°C), cough, dyspnea, myalgia and fatigue, respiratory symptoms, gastrointestinal symptoms (such as diarrhea) within 7 days prior to the hospital stay (all periods);
* Having had direct and significant contact, at the medical discretion, with people who tested positive for a coronavirus test within 14 days prior to the hospital stay (all periods);
* Living in the same household as people who fall into the risk group of worse prognosis for coronavirus infection, such as individuals over 60 years old, individuals with respiratory problems, immunosuppressed or those with chronic diseases such as heart or diabetes (all periods );
* Any clinical condition or laboratory alteration that, at the investigator's discretion, may compromise trial participation, ie:
* Have an abnormal erythrocyte count (<4.0 M/mm3 or >5.4 M/mm3);
* Have an abnormal reticulocyte count (> 3.0%);
* Have an abnormal platelet count (< 135,000/μL or > 550,000/μL);
* Have an abnormal hemoglobin level (< 13g/dL);
* Have an abnormal level of hematocrit (<40% or >54%);
* Have an abnormal level of ferritin (< 100 ng/mL or > 336.2 ng/mL);
* Have an abnormal level of transferrin (< 200 mg/dL or > 360 mg/dL);
* Have an abnormal level of transferrin saturation (<20%)
* Have abnormal levels of vitamin B12 (< 130 pg/mL or >868 pg/mL);
* Present evidence of cardiovascular disorders, particularly arterial hypertension (supine blood pressure > 145 / 90mmHg at baseline);
* History of venous thrombosis;
* Participants diagnosed with iron deficiency anemia or clinical history of autoimmune or hereditary anemia;
* Clinical history of chronic or acute hemorrhages in the 30 days preceding the start of the trial;

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-06 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of AUC0-inf | 14 days
  Area under curve Cp(t) rHuEpo from time zero to infinity
Evaluation Cmax | 14 days
  Maximum plasma concentration for rHuEpo
Evaluation of Emax | 14 days
  maximum increase in reticulocyte count
Evaluation of ASEC0-t | 14 days
  Area under curve reticulocyte count f(t) from time zero to day 14

SECONDARY OUTCOMES:
half life | 14 days
  Compare profiles for T½ between the experimental drug and the comparator.
Tmax | 14 days
  Compare profiles for Tmax between the experimental drug and the comparator.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Kumar, MD, Principal Investigator — Azidus Principal Investigator
Locations (1):
- Azidus Laboratories, Chennai, India